CLINICAL TRIAL: NCT01460459
Title: Self-monitoring of Blood Glucose in Insulin-treated Patients With Type 2 Diabetes: a 9-month Randomised Controlled Trial
Brief Title: Self-monitoring of Blood Glucose in Insulin-treated Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Foundation, The Netherlands (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35308.075.11
Record Dates: First submitted 2011-10-19; First posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; self-monitoring of blood glucose; frequency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- high frequency of SMBG (Experimental): Patients are instructed to measure their blood glucose concentrations 4 times per day (pre-prandial and before bedtime) one day weekly in group A.
  Interventions: Behavioral: a specific frequency of SMBG
- middle frequency of SMBG (Experimental): Patients are instructed to measure their blood glucose concentrations 4 times per day (pre-prandial and before bedtime) one day per two weeks in group B.
  Interventions: Behavioral: a specific frequency of SMBG
- low frequency of SMBG (Experimental): Patients are instructed to measure their blood glucose concentrations 4 times per day (pre-prandial and before bedtime) Group C: one day monthly
  Interventions: Behavioral: a specific frequency of SMBG

INTERVENTIONS:
Behavioral: a specific frequency of SMBG — Patients are instructed to measure their blood glucose concentrations 4 times per day (pre-prandial and before bedtime:
  high frequency: one day weekly middle frequency:one day per two weeks low frequency:one day monthly

SUMMARY:
Primary Objective:

The objective of the study is to investigate the effect of a specific frequency of Self-monitoring of blood glucose (SMBG) on glycemic control and quality of life in patients with type 2 diabetes and who are in stable good glycemic control and using 1 insulin injection daily.

The research question is:

Does a less intensive frequency of SMBG in insulin-treated patients with type 2 diabetes, who are in stable good glycemic control, using 1 insulin injection daily, lead to a clinically relevant increase of HbA1c (an increase of 0.5%) and what is the effect on quality of life?

Secondary objectives:

The secondary objectives is to investigate the effect of a specific frequency of SMBG on the number of hypo and hyper glycaemia, number of extra diabetes-related contacts with the health care provider, and the diabetes medication.

DETAILED DESCRIPTION:
SUMMARY

Rationale:

Self-monitoring of blood glucose (SMBG) is an important tool in diabetes care to achieve and maintain good glycemic control. But how often 'should' the patient measure the capillary glucose concentration? There is no general agreement between professionals, and there is no evidence for a specific frequency and timing.

Objective:

The objective of the study is to investigate the effect of a specific frequency of SMBG on glycemic control and quality of life in patients with type 2 diabetes and who are in stable good glycemic control and using 1 insulin injection daily.

Study design:

An open Randomised Controlled Trial.

Study population:

Patients with insulin-treated diabetes type 2, > 18 years of age, using 1 insulin injection daily, performing SMBG > 1 year, HbA1c ≤ 58 mmol/mol (< 7.5%) in the preceding 12 months, sufficient knowledge of the Dutch language, no hypo-unawareness, no serious co-morbidity

Intervention:

Patients are instructed to measure their blood glucose concentrations 4 times per day (pre-prandial and before bedtime) one day weekly in group A, one day per two weeks in group B and one day monthly in group C. Patients are asked to keep a diary with the readings and the probably extra measurements, including the reasons.

Main study parameters/endpoints:

The main study parameters are glycemic control and quality of life. A difference of > 0.5% (> 5.5 mmol/mol) in HbA1c is considered to be relevant. Quality of life is measured with 3 validated questionnaires.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients in this study are used to perform SMBG. During the study, they are asked to monitor their glucose concentrations in a controlled, specific frequency (different kind of usual care are compared). And they are asked to fill in 3 questionnaires in the beginning and at the end of the study. Extra HbA1c measurements can be necessary. No side effects are expected, but safety is incorporated through HbA1c measurements every 3 months and every 3 months the diary will be discussed in the scheduled visits. Furthermore, extra measurements are allowed when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients with insulin-treated diabetes type 2
* > 18 years of age
* using 1 insulin injection daily,
* performing SMBG > 1 year
* HbA1c ≤ 58 mmol/mol (< 7.5%) in the preceding 12 months
* sufficient knowledge of the Dutch language.-

Exclusion Criteria:

* no hypo-unawareness
* no serious co-morbidity (as judged by their own GP)
* patients who measure their blood glucose concentration (4 measurements a day) more than once a week on average

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 9 months
  The main study parameter is glycemic control. Glycemic control is measured by HbA1c. A difference of 0.5% (> 5.5 mmol/mol) in HbA1c between groups is considered to be relevant.

SECONDARY OUTCOMES:
quality of life | 9 months
  The secondary study parameter is quality of life. The quality of life is measured by 3 validated questionnaires: the 12-item Short Form Health Survey, the 20-item Problems Areas in Diabetes Scale (PAID) and the 13-item Summary of Diabetes Self care Activities. Furthermore, the glucose concentrations measured by SMBG should be between 4-7 mmol/l, preprandial and between 8-10 mmol/l before bed time. The endpoint is the number of glucose concentrations who are out of range at every 4th week.The number of hypo and hyperglycaemia are reported in the diary.

CONTACTS AND LOCATIONS:
Overall Officials: Henk JG Bilo, MD PhD FCRP, Principal Investigator — Isala
Locations (1):
- Diabetes Centre, Isala Clinics, Zwolle, Netherlands

REFERENCES:
- [Derived] Hortensius J, Kleefstra N, Landman GWD, Houweling BT, Groenier KH, van der Bijl JJ, Bilo H. Effects of three frequencies of self-monitored blood glucose on HbA1c and quality of life in patients with type 2 diabetes with once daily insulin and stable control: a randomized trial. BMC Res Notes. 2018 Jan 15;11(1):26. doi: 10.1186/s13104-018-3138-7. PMID 29334997